CLINICAL TRIAL: NCT01433393
Title: Double-blind Comparative Study of TAK-875
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Model: Parallel
Other Study IDs: TAK-875/CCT-003; U1111-1124-1518 (Registry Identifier: WHO); JapicCTI-111604 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus | interventions — TAK-875

ARMS (3):
- TAK-875 25 mg (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 50 mg (Experimental)
  Interventions: Drug: TAK-875
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-875
  Arms: TAK-875 25 mg
Drug: TAK-875
  Arms: TAK-875 50 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treatment with TAK-875 in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is an outpatient.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. The participant has any serious cardiac disease, serious cerebrovascular disorder, or any serious pancreatic or hematological disease.
2. The participant is considered ineligible for the study for any other reason by the investigator or sub-investigator.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HbA1c

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Kisarazu-shi, Chiba
  - Matsuyama, Ehime
  - Fukuoka-shi Nishi-ku, Fukuoka
  - Kasuga-shi, Fukuoka
  - Naka, Ibaragi
  - Tsuchiura-shi, Ibaragi
  - Takamatsu, Kagawa-ken
  - Kyoto-shi Fushimi-ku, Kyoto
  - Nagasaki, Nagasaki
  - Kashihara-shi, Nara
  - Kashiwara-shi, Osaka
  - Osaka-shi Tsurumi-ku, Osaka
  - Sakai-shi Nishi-ku, Osaka
  - Shimotsuke-shi, Tochigi
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toshima-ku, Tokyo